CLINICAL TRIAL: NCT07341503
Title: The Sleep After Breast Cancer (ABC) Study - Examining Sleep Changes and Biomarkers Among Breast Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: American Association for Cancer Research (Other)
Responsible Party: Principal Investigator, Electra Paskett, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-24386; NCI-2025-02354 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-09-18; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-09

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Breast Carcinoma; Hormone Receptor-Positive Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cheek swab, saliva, and hair samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients undergo collection of cheek swab, saliva, and hair samples, wear a wrist sleep tracking device, and complete surveys throughout the study. Additionally, patients have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study
  Other Names: Non-Interventional Observational Study; Noninterventional (Observational) Study

SUMMARY:
This study is being done to learn more about breast cancer patients' experiences with sleep changes during cancer treatment, identify possible reasons for poor sleep quality, and to find out how stress, social support, and living environment affect sleep.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Characterize longitudinal trends in sleep among BC patients from treatment through survivorship, overall and by race, ethnicity, and underserved communities (rural, urban, Appalachian) using actigraphy-assessed sleep duration (Aim 1a), and self-reported sleep quality (Aim 1b).

II. Identify risk factors (sociodemographic, clinical treatment, social support, built environment) associated with sleep duration and sleep quality over time.

III. Assess how sleep duration and quality affect premature biological aging, stress, and inflammatory markers in BC patients from treatment to survivorship, overall and by race, ethnicity, and community.

OUTLINE: This is an observational study.

Patients undergo collection of cheek swab, saliva, and hair samples, wear a wrist sleep tracking device, and complete surveys throughout the study. Additionally, patients have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* * Age >= 18 years old at time of breast cancer diagnosis

  * Stage I to III breast cancer diagnosis
  * Hormone receptor positive breast cancers
  * Post primary surgery, before chemotherapy/radiation therapy begins
  * No known evidence of breast cancer recurrence (local or distant) or second, primary cancer
  * No prior history of new other malignancy since their breast cancer diagnosis (other than non-melanoma skin cancer)
  * Able to speak, understand and read English
  * Cognitively able to complete the study requirements
  * Ability to access medical records from treating hospital

Exclusion Criteria:

* * Stage IV or metastatic breast cancer

  * Not cognitively able to provide informed consent
  * Not willing to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with stage I to stage III breast cancer, being followed at the OSUCCC.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total sleep duration | Through study completion, an average of 9 months
  Will report descriptive statistics of the sample characteristics using counts and percentages or means and standard deviations. Actigraphy from the sleep watch (GENEActiv device) will be scored and analyzed using validated algorithms within the Activeinsights software (Activinsights, UK). Daily and weekly summaries of sleep statistics will be averaged to generate person-level data for analysis at each time point. a paired t-test to compare T1 sleep duration (pre-treatment) to T3 (treatment completion) sleep duration using SAS PROC POWER.
Self-reported sleep quality (PROMIS) | Through study completion, an average of 9 months
  Sleep quality (as measured by the PROMIS) will be considered as a continuous variable and categorized into 'poor quality' if patients have a score of >= 5 and 'good quality' if < 5 points. Locally weighted scatterplot smoothing will be used to estimate a smooth trend through the sleep data points (sleep duration, sleep quality). Generalized linear mixed models will be used to examine changes in sleep over time (treatment through survivorship).

CONTACTS AND LOCATIONS:
Overall Officials: Electra Paskett, MSPH, PhD, FAACR, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States